CLINICAL TRIAL: NCT03513276
Title: Effect of Local Infiltration Anesthesia in a Hip Arthroplasty Fast Track Program.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, fangles, Medical Doctor, Hospital Mutua de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00002
Record Dates: First submitted 2018-02-26; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Saline Solution; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Multimodal analgesia + Local Infiltration Anesthesia (Experimental): 100cc of 2% ropivacaine + Adrenaline 10mcg/ml + 20cc saline solution
  Interventions: Drug: 100cc of 2% ropivacaine; Drug: Adrenaline 10mcg/ml
- Multimodal analgesia + saline solution (Active Comparator): 120cc of saline solution
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: 100cc of 2% ropivacaine — Multimodal analgesia + Local infiltration anesthesia
  Arms: Multimodal analgesia + Local Infiltration Anesthesia
Drug: Saline Solution — Multimodal analgesia + Saline solution
  Arms: Multimodal analgesia + saline solution
Drug: Adrenaline 10mcg/ml
  Arms: Multimodal analgesia + Local Infiltration Anesthesia

SUMMARY:
Fast-track programs in Orthopaedic Surgery require early motion that can only be achieved by optimal pain management protocols. Multimodal analgesia protocols including local infiltration anesthesia (LIA) have obtained excellent results in fast-track programs involving Total Knee Arthroplasty but further research and data is needed in Total Hip Arthoplasty programs.

ELIGIBILITY:
Inclusion Criteria:

* Hip osteoarthritis requiring Total Hip Replacement

Exclusion Criteria:

* Mental Disorders
* contraindications for epidural anesthesia
* Neurologic disorders that could interfere with pain evaluation
* allergy to drugs in multimodal analgesic protocol

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Pain measured in Visual Analog Scale | Up to 48h postoperatively
  Pain assesed using Visual Analog Scale ( Scoring from 0 to 10)

SECONDARY OUTCOMES:
Length of hospital stay | Up to 1 week
  Length of hospital stay measured in days
Analgesic requirements | Up to 1 week
  Analgesia requirements needed besides protocol medication Measured in miligrams of drug required(Sevredol) Analgesia required by patient
Complications | Up to 1 week
  Wound dehiscence, Infection, reoperation, dislocation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Derived] Bernaus M, Novellas M, Bartra A, Nunez JH, Angles F. Local infiltration analgesia does not have benefits in fast-track hip arthroplasty programmes: a double-blind, randomised, placebo-controlled, clinical trial. Hip Int. 2022 Nov;32(6):711-716. doi: 10.1177/1120700021992684. Epub 2021 Feb 18. PMID 33601948